CLINICAL TRIAL: NCT05198518
Title: Utilization of a Microcurrent Device for Postoperative Pain Following Functional Endoscopic Sinus Surgery: a Randomized Controlled Trial
Brief Title: Microcurrent Device (TIVIC Health)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Tivic Health Systems (Industry)
Responsible Party: Principal Investigator, Alfred-Marc Iloreta, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-21-01392
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Chronic Rhinosinusitis
Keywords: chronic rhinosinusitis; postoperative pain; microcurrent
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned in a 1:1 ratio to receive the intervention or placebo. Randomization will be completed via a computer-generated randomization table.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant and all study staff will be blinded to which device they are receiving, either the study device or the identical sham device. Devices will be labeled A or B, with only the device manufacturer knowing which device is the active study device and which is the sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Microcurrent TENS device (Experimental): A handheld micro-current TENS emitter device, which applies a small current of electricity to the forehead and maxillary region
  Interventions: Device: Microcurrent TENS device
- Sham device (Sham Comparator): The sham device appears identical to the active device while emitting no therapeutic microcurrent.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Microcurrent TENS device — The study device is a handheld micro-current TENS emitter intended to be used for the relief of postoperative pain after FESS. The design of the study device was optimized to provide transcutaneous nerve stimulation to the regional areas associated with the sinuses.
  Other Names: Microcurrent neuromodulation device
  Arms: Microcurrent TENS device
Device: Sham Device — The sham device appears and operates identically to the active device, including indicator lights and haptic vibration, however it emits a weak direct current that is non-therapeutic.
  Arms: Sham device

SUMMARY:
The purpose of this study is to investigate whether daily use of a microcurrent neuromodulation device, which applies a small current of electricity to the forehead and maxillary region, will decrease the pain experienced by patients in the days following functional endoscopic sinus surgery (FESS). This study is a prospective randomized controlled study. Enrolled subjects will be randomized (1:1) to receive either an active neuromodulation study device or a sham device that appears identical to the active device while emitting no therapeutic microcurrent. Subjects will self-treat with the device at home and will be followed for 2 weeks after FESS.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for FESS functional nasal or endoscopic sinus surgery
* Possessing an American Society of Anesthesiologists physical status classification of I or II
* Age ≥ 18
* Possess the capacity to give informed consent
* Able to read, write and understand English or Spanish
* Able to attend follow up visits at postop days 7 and 14 Visit 1 (within 0 - day 14) and post-op Visit 2 (within 10 - 21 days)
* Postop pain VAS ≥ 5 in PACU phase II

Exclusion Criteria:

* Age < 18
* Does not understand English or Spanish
* Does not meet inclusion criteria
* History of chronic pain
* Experiencing chronic pain requiring opioids at baseline and/or who are under the care of pain management specialists
* Neurologic disorders (including seizure disorders)
* Undergoing planned or unplanned additional procedures at the time of FESS surgery
* In custody of the state
* Prisoners
* Known to be pregnant
* Implanted cranial metallic components or devices including deep brain stimulators or cochlear implants
* Has an implanted or external worn cardiac device including pacemakers, automated implantable cardioverter defibrillator (AICD), or any other cardiac electric devices (including non-implanted devices, e.g. defibrillator vest)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred-Marc Iloreta, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Faculty Practice Associates - Mount Sinai Doctors, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No additional clinically relevant information will be collected from subjects in the course of the study beyond what is routinely collected and communicated to patients in their standard course of care. Study subjects will not be notified of results until the final analysis of study data is complete. The study results will be submitted for publication and/or presentation at national conferences/journals.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 patients met the inclusion criteria and enrolled into the study.
Groups:
- All Participants Screened: Participants consented and had screening visit to determine eligibility
Period: Screening Visit
Arm/Group | All Participants Screened | Microcurrent TENS Device | Sham Device
Started | 118 | 0 | 0
Completed | 60 | 0 | 0
Not Completed | 58 | 0 | 0
Not completed — Deemed unable to participate | 58 | 0 | 0
Period: Enrolled Participants
Arm/Group | All Participants Screened | Microcurrent TENS Device | Sham Device
Started | 0 | 27 | 33
Completed | 0 | 27 | 33
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Microcurrent TENS Device | Sham Device | Total
Number analyzed (Participants) | 27 | 33 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.38 (14.63) | 39.55 (14.31) | 40.35 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 17 | 23 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (Caucasian) | 19 | 17 | 36
  Black or African American | 4 | 6 | 10
  Hispanic or Latino | 2 | 5 | 7
  Asian | 0 | 3 | 3
  Other | 0 | 1 | 1
Prior Sinus Surgery [Count of Participants; unit: Participants] | 25 | 5 | 30
Pre-Operative Diagnosis [Count of Participants; unit: Participants]
  Chronic Rhinosinusitis without Polyposis | 16 | 19 | 35
  Chronic Rhinosinusitis with Polyposis | 8 | 6 | 14
  Other | 3 | 8 | 11
Septoplasty [Count of Participants; unit: Participants] | 18 | 22 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Visual Analog Score After First Use of Device
Description: Change in postoperative pain score in first use of device post-op at different timepoints after intervention. Participants will record their pain score before and after use of the device. The pain will be recorded using a visual analog scale. Full scale from 0-10, with higher score indicating more pain.
  Participants instructed to use device for total of 14 days and recommended to use at least 3x a day. They are asked to record their pain levels at baseline, 10 min, 2 hours, and 4 hours after the first time they use the device.
Time Frame: baseline, 10 min, 2 hour, 4 hour at first use within 14 days after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 4.9 (2.06) | 5.6 (2.68)
  10 min | 4.7 (1.96) | 4.8 (2.31)
  2 hour | 4.0 (2.26) | 4.2 (2.33)
  4 hour | 3.7 (2.47) | 3.9 (2.46)

2. Primary Outcome: Change in Pain Visual Analog Score After Second Use of Device
Description: Change in postoperative pain score after second use of device post-op at different timepoints after intervention. Participants will record their pain score before and after use of the device. The pain will be recorded using a visual analog scale. Full scale from 0-10, with higher score indicating more pain.
  Participants instructed to use device for total of 14 days and recommended to use at least 3x a day. They are asked to record their pain levels at baseline, 10 min, 2 hours, and 4 hours after the second time they use the device.
Time Frame: baseline, 10 min, 2 hour, 4 hour at second use within 14 days after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 4.4 (1.91) | 5.7 (2.99)
  10 min | 3.8 (1.60) | 5.0 (2.62)
  2 hour | 3.6 (1.66) | 4.5 (2.56)
  4 hour | 3.6 (1.66) | 4.2 (2.11)

3. Primary Outcome: Change in Pain Visual Analog Score After Third Use of Device
Description: Change in postoperative pain score after third use of device post-op at different timepoints after intervention. Participants will record their pain score before and after use of the device. The pain will be recorded using a visual analog scale. Full scale from 0-10, with higher score indicating more pain.
  Participants instructed to use device for total of 14 days and recommended to use at least 3x a day. They are asked to record their pain levels at baseline, 10 min, 2 hours, and 4 hours after the third time they use the device.
Time Frame: baseline, 10 min, 2 hour, 4 hour at 3rd use within 14 days after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 4.7 (2.20) | 4.6 (3.05)
  10 min | 4.3 (2.20) | 4.3 (2.47)
  2 hour | 3.6 (2.02) | 4.0 (1.84)
  4 hour | 3.7 (2.09) | 3.8 (2.07)

4. Primary Outcome: Change in Pain Visual Analog Score After Fourth Use of Device
Description: Change in postoperative pain score after fourth use of device post-op at different timepoints after intervention. Participants will record their pain score before and after use of the device. The pain will be recorded using a visual analog scale. Full scale from 0-10, with higher score indicating more pain.
  Participants instructed to use device for total of 14 days and recommended to use at least 3x a day. They are asked to record their pain levels at baseline, 10 min, 2 hours, and 4 hours after the fourth time they use the device.
Time Frame: baseline, 10 min, 2 hour, 4 hour at fourth use within 14 days after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 4.4 (2.06) | 4.1 (2.48)
  10 min | 3.6 (1.96) | 4.1 (2.35)
  2 hour | 3.3 (1.84) | 3.5 (2.15)
  4 hour | 3.1 (1.85) | 3.3 (2.22)

5. Primary Outcome: Change in Pain Visual Analog Score After Fifth Use of Device
Description: Change in postoperative pain score after fifth use of device post-op at different timepoints after intervention. Participants will record their pain score before and after use of the device. The pain will be recorded using a visual analog scale. Full scale from 0-10, with higher score indicating more pain.
  Participants instructed to use device for total of 14 days and recommended to use at least 3x a day. They are asked to record their pain levels at baseline, 10 min, 2 hours, and 4 hours after the fifth time they use the device.
Time Frame: baseline, 10 min, 2 hour, 4 hour at fifth use within 14 days after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 3.6 (1.71) | 4.1 (2.70)
  10 min | 3.3 (1.50) | 3.8 (2.48)
  2 hour | 3.4 (1.51) | 2.9 (2.02)
  4 hour | 2.9 (1.31) | 2.7 (2.28)

6. Primary Outcome: Sino-Nasal Outcome Test (SNOT 22)
Description: The possible range of Total SNOT scores is between 0 to 110. Higher scores indicate greater rhinosinusitis-related health burden.
Time Frame: Baseline and 2 weeks Post-Op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 46.5 (21.4) | 37.6 (21.8)
  2 weeks post-op | 27.0 (17.5) | 19.2 (15.9)

7. Primary Outcome: Mean Difference in Nasal Obstruction Symptom Evaluation (NOSE) Score
Description: Full scale from 0-100. Higher score indicates more severe symptoms
Time Frame: Baseline and 2 weeks Post-Op
Measure: Mean (Standard Deviation); unit: mean difference in score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
mean difference in score on a scale | 3.8 (4.8) | 3.8 (7.4)

8. Secondary Outcome: Debridement Associated Pain Visual Analog Score Before Use of Device
Description: Participants will record their pain before using the device at their postoperative debridement visits on post operative day 14 (POD14). Their pain levels will be recorded at baseline, 10 min, 2 hours, and 4 hours using a visual analog scale. Full scale from 0-10, with higher score indicating more pain.
Time Frame: baseline, 10 min, 2 hour, 4 hour on POD14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 4.88 (2.06) | 5.6 (2.68)
  10 min | 4.71 (1.96) | 4.8 (2.31)
  2 hour | 4 (2.26) | 4.2 (2.33)
  4 hour | 3.71 (2.47) | 3.85 (2.46)

9. Secondary Outcome: Debridement Associated Pain Visual Analog Score After First Use of Device
Description: Participants will record their pain before using the device at their postoperative debridement visits on post operative day 14 (POD14). Their pain levels will be recorded at baseline, 10 min, 2 hours, and 4 hours after the first use of device using a visual analog scale. Full scale from 0-10, with higher score indicating more pain.
Time Frame: baseline, 10 min, 2 hour, 4 hour on POD14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 4.47 (1.91) | 5.67 (2.99)
  10 min | 3.76 (1.6) | 5 (2.62)
  2 hour | 3.59 (1.66) | 4.53 (2.56)
  4 hour | 3.59 (1.66) | 4.2 (2.11)

10. Secondary Outcome: Debridement Associated Pain Visual Analog Score After Second Use of Device
Description: Participants will record their pain before using the device at their postoperative debridement visits on post operative day 14 (POD14). Their pain levels will be recorded at baseline, 10 min, 2 hours, and 4 hours after the second use of device using a visual analog scale. Full scale from 0-10, with higher score indicating more pain.
Time Frame: baseline, 10 min, 2 hour, 4 hour on POD14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 4.71 (2.2) | 4.6 (3.05)
  10 min | 4.29 (2.2) | 4.25 (2.47)
  2 hour | 1.82 (3.64) | 2.02 (4)
  4 hour | 3.71 (2.09) | 3.8 (2.07)

11. Secondary Outcome: Debridement Associated Pain Visual Analog Score After Third Use of Device
Description: Participants will record their pain before using the device at their postoperative debridement visits on post operative day 14 (POD14). Their pain levels will be recorded at baseline, 10 min, 2 hours, and 4 hours after the third use of device using a visual analog scale. Full scale from 0-10, with higher score indicating more pain.
Time Frame: baseline, 10 min, 2 hour, 4 hour on POD14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 4.4 (2.06) | 4.06 (2.48)
  10 min | 3.6 (1.96) | 4.11 (2.35)
  2 hour | 3.33 (1.84) | 3.5 (2.15)
  4 hour | 3.13 (1.85) | 3.33 (2.22)

12. Secondary Outcome: Debridement Associated Pain Visual Analog Score After Fourth Use of Device
Description: Participants will record their pain before using the device at their postoperative debridement visits on post operative day 14 (POD14). Their pain levels will be recorded at baseline, 10 min, 2 hours, and 4 hours after the fourth use of device using a visual analog scale. Full scale from 0-10, with higher score indicating more pain.
Time Frame: baseline, 10 min, 2 hour, 4 hour on POD14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
score on a scale
  Baseline | 3.75 (1.71) | 4.13 (2.7)
  10 min | 3.33 (1.5) | 3.8 (2.48)
  2 hour | 3.41 (1.51) | 2.93 (2.02)
  4 hour | 2.91 (1.31) | 2.73 (2.28)

13. Secondary Outcome: Postoperative Pain Medication Usage
Description: Participants will record their postoperative pain medication daily usage (opioids and acetaminophen). Number of Acetaminophen 325mg or Number of Oxycodone 5 mg taken across 2 weeks post-op
Time Frame: Daily until 2nd postoperative visit (day 14)
Measure: Mean (Standard Deviation); unit: number of pills
Arm/Group | Microcurrent TENS Device | Sham Device
Number analyzed (Participants) | 27 | 33
number of pills
  Tylenol | 24.3 (30.83) | 16.4 (14.87)
  Oxy | 2.5 (2.84) | 1.5 (2.29)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Microcurrent TENS Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/33
Other Adverse Events (participants affected / at risk) | 0/27 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT05198518/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT05198518/ICF_001.pdf